CLINICAL TRIAL: NCT07205965
Title: The Effect of Acceptance and Commitment Therapy-Based Psychoeducation on Anxiety, Depressive Symptoms, Psychological Flexibility, Mindfulness and Valuing in Cancer Survivors: A Randomized Controlled Trials
Brief Title: The Effect of Acceptance and Commitment Approach-Based Psychoeducation in Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Neslihan Partlak Günüşen, Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8122-GOA
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Cancer Breast; Colon Cancer; Cancer Survivors
Keywords: depression; anxiety; Mindfulness; Values; Acceptance and commitment approach; Psychological flexibility; cancer survivor
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The control group will not receive any intervention during the application period and will be put on waitlist.
- experimental/group (Experimental): The experimental group will consist of 16 participants and the participants will receive internet-based environment psychoeducation for 6 weeks, each session for 30 minutes.
  Interventions: Behavioral: Experimental Group

INTERVENTIONS:
Behavioral: Experimental Group — The experimental group will consist of 16 participants and the participants will receive internet-based environment psychoeducation for 6 weeks, each session for 30 minutes.
  Arms: experimental/group

SUMMARY:
The study is planned to be conducted in a randomised controlled experimental design in accordance with CONSORT. The study is planned to be conducted between September 2025 and December 2026 at X Hospital with individuals who have completed cancer treatment. The randomisation list will be concealed from the participants, and each participant will be informed of which group they have been assigned to after being included in the study. The 'Stratified Randomisation' method will be used to determine which group participants will be assigned to, and participants will be included in the study based on their scores on the HAD scale. They will then be divided into experimental and control groups. To prevent study bias, the assignment of intervention and control groups will be conducted by an expert who has not participated in the study, with the aim of keeping the randomisation information confidential. The experimental group will consist of a total of 16 participants and will receive individual psychoeducation in an internet-based environment for 6 weeks, with each session lasting 30 minutes. No intervention will be made to the control group during the application period, and they will be placed on a waiting list. Participants who complete the psychoeducation will undergo follow-up measurements via an internet-based platform one month, six months, and one year after the psychoeducation, and their scores will be compared with those of the control group. The sample criteria include: having completed cancer treatment, having completed treatment for breast, gynaecological, colon or rectal cancer, having internet access, and being at risk for depression or anxiety in one or both of these sub-dimensions according to the Hospital Anxiety and Depression (HAD) scale. Exclusion criteria include receiving another psychosocial intervention, using psychiatric medication other than antidepressants, being in an advanced stage of cancer, having metastatic cancer, having recurrent cancer, and having started antidepressants in the last three months. Participants will be asked to complete a demographic information form. In addition, anxiety and depression levels will be measured using the Hospital Anxiety and Depression (HAD) scale. Psychological flexibility will be measured using the Acceptance and Action Questionnaire-II, mindfulness will be measured using the Mindfull Attention Awareness Scale, and the level of valuing will be measured using the Valuing Questionnaire. Validity and reliability studies have been conducted for the scales. Ethical committee approval has been obtained. Institutional approval has been obtained from the hospital where the study is being conducted.

DETAILED DESCRIPTION:
According to World Health Organisation data, approximately one in six deaths is due to cancer (WHO, 2022). With the development of healthcare services, cancer survival rates are increasing and progress is being made in the treatment of the disease, but the physical and psychosocial effects of cancer on individuals continue (Li, Guo, Li & Yang, 2021). In recent years, new approaches have been developed to support the mental well-being of cancer patients. The foremost of these is Acceptance and Commitment Therapy (ACT). ACT is an approach developed as a result of the interaction between empirical data obtained from scientific research on human behaviour and clinical experience. ACT, which comes from a humanistic model, emphasises awareness and self-compassion. As a behavioural therapy, ACT draws its origins from the perspectives of Skinner and Pavlov and is based on the Relational Frame Theory, which focuses on the nature of human language and cognitive processes. ACT aims to increase functionality and enable individuals to live more meaningful and valuable lives by using mindfulness. ACT intervention consists of six important cognitive processes. These are a therapeutic approach model consisting of values, contact with the present moment, cognitive defusion, acceptance, contextual self, and committed action. The aim of this study is to examine the effect of acceptance and commitment therapy-based psychoeducation applied to cancer survivors on individuals' anxiety, depressive symptoms, psychological flexibility, acceptance, value-oriented life, and awareness.

The study consists of survivors diagnosed with one of the following types of cancer: breast, gynaecological, colon, or rectal. Participants will be invited to join the study via telephone from the oncology unit's database, targeting patients who have completed these treatments within the past 1-12 months. Accepting patients will first be interviewed in person, and the HAD scale will be administered. Participants who meet the eligibility criteria will be included in the study. Inclusion criteria: - Being between 18 and 65 years of age, having completed cancer treatment, being able to speak Turkish, and, according to the Hospital Anxiety and Depression (HAD) scale, having distress in one or both of the depression or anxiety subscales (HAD-A ≥ 10 and/or HAD-D ≥ 7 based on the cut-off score), and having internet access. The exclusion criteria for the study are receiving another psychosocial intervention, cancer metastasis or recurrence, use of psychiatric medication other than antidepressants, and initiation of antidepressant treatment in the last three months.

The aim of this study is to examine the effect of acceptance and commitment therapy-based psychoeducation applied to cancer survivors on individuals' anxiety, depressive symptoms, psychological flexibility, acceptance, value-oriented life, and awareness.

For the sample calculation required for the study, the G power statistical analysis programme was used, with a Type I error of 0.05, a Type II error of 0.20 (power 0.80), and an effect size of 0.25, and an ANOVA test was applied. Anticipating possible losses in the sample, a total of 32 participants, 16 in each group, are planned to be included. In the data analysis of the study, descriptive statistics will be expressed as numbers (n) and percentages (%) for discrete variables and as mean ± standard deviation (minimum-maximum) for continuous variables. In all analyses, p-values less than 0.05 will be considered statistically significant. The normality of continuous variables will be determined based on Shapiro-Wilks test values, normality tests, and histograms. The similarity of the experimental and control groups will be evaluated using the chi-square test for categorical variables and the t-test for continuous variables. The comparison of the levels of the outcome variables of the experimental and control groups before the intervention will be performed using the t-test. For the evaluation of repeated measurements (depressive symptoms, psychological flexibility, mindfulness, and value), a two-way analysis of variance will be used. For the evaluation of missing data, the Intention to Treat principle will be applied.

The study is planned to be conducted in a randomised controlled experimental design in accordance with CONSORT. The study is planned to be conducted between September 2025 and December 2026 at X Hospital with individuals who have completed cancer treatment. Individuals who are at risk for depression or anxiety in one or both of these sub-dimensions according to the Hospital Anxiety and Depression (HAD) scale will participate in the study. Individuals will be contacted by telephone and will first undergo a face-to-face interview. The psychoeducation sessions will be conducted online, individually, in approximately 30-minute sessions over 6 sessions. A total of 32 individuals will be included in the study, with 16 in the experimental group and 16 in the control group. Follow-ups will be conducted before the intervention, after the intervention, at 3 months, 6 months, and 12 months. No intervention will be performed on the control group during the application period, and they will be placed on a waiting list. If the intervention is found to be effective after the study is completed, it is planned to apply the programme to the volunteer participants in the control group.

The randomisation list will be concealed from participants, and each participant will be informed of their group assignment after being included in the study. Participants will be assigned to the experimental and control groups using the 'stratified randomisation' method based on their scores to determine which group they will be included in. To prevent study bias, the assignment of participants to the intervention and control groups will be conducted by an expert who is not involved in the study, in order to conceal the random assignment information.

In the study, participants will be asked to complete a demographic information form. Anxiety and depression levels will be measured using the Hospital Anxiety and Depression Scale (HADS). Psychological flexibility will be measured using the Acceptance and Action Questionnaire-II, mindfulness will be measured using the Mindfull Attention Awareness Scale, and the level of valuing will be measured using the Valuing Questionnaire. The validity and reliability of the scales have been established. Institutional permission has been obtained from the hospital where the study is being conducted. The study has been approved by the ethics committee of the relevant university. Additionally, verbal and written consent will be obtained from participants; individuals will be informed that information about them will not be shared with others and that the 'principle of confidentiality' will be adhered to. The costs of the study will be covered by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* having completed cancer treatment, having completed treatment for breast, gynaecological, colon or rectal cancer, having internet access, and being at risk for depression or anxiety in one or both of these sub-dimensions according to the Hospital Anxiety and Depression (HAD) scale.

Exclusion Criteria:

* receiving another psychosocial intervention, using psychiatric medication other than antidepressants, being in an advanced stage of cancer, having metastatic cancer, having recurrent cancer, and having started antidepressants in the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Change from to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention.
  The Hospital Anxiety and Depression Scale (HADS) is used to measure participants' anxiety and depression levels. In this scale (HADS), there are seven questions each to measure the dimensions of depression and anxiety. Each subscale consists of seven items with a 4-point ordinal response format. Scores ranges from 0 to 21 in each subscale, with higher scores indicating higher levels of anxious or depressive state. The scale has a four-point Likert-type. The cut-off points for the Turkish form of the HADS Scale are 10 for the anxiety subscale (HAD-A) and 7 for the depression subscale (HAD-D).

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire-II (AAQ-II) | Change from baseline psychological flexibility levels to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention.
  The seven-item Acceptance and Action Questionnaire-II is a reliable and valid scale for measuring psychological flexibility in both clinical and non-clinical samples. The mean Cronbach Alpha coefficient was found to be .84, and the internal consistency was high.The questionnaire consists of seven items in total. The scale items are graded from 1 (never true) to 7 (always true). The lowest score to be taken from the scale is 7 and the highest score is 49. The AAQ-II is a seven-point Likert-type scale, and as the total score increases, psychological rigidity increases and psychological flexibility decreases.
Mindful Attention Awareness Scale (MAAS) | Change from baseline mindfulness levels to the end point of the intervention and one month (4 weeks), six months (24 weeks), 12 months (48 weeks) after the intervention.
  Mindful Attention Awareness Scale was developed to measure the general level of mindfulness and attention to current processes in daily life. The Cronbach Alpha internal consistency coefficient calculated for the reliability of the scale is 0.80. The scale consists of 15 items. The lowest score that can be obtained from the scale is 15 and the highest 90. The scale is a 6-point Likert type scale: almost always (1), often (2), sometimes (3), rarely (4), rarely (5), almost never (6). The Mindful Attention Awareness Scale has a single factor and a single total score is obtained from the scale. As the score obtained from the scale increases, the level of mindfullness of the individual increases.
The Valuing Questionnaire | Change from baseline valuing levels to the end point of the intervention and one month (4 weeks), six months (2.4 weeks), 12 months (48 weeks) after the intervention
  The Valuing Questionnaire measures the extent to which people live in accordance with the value they have determined in the last week. The questionnaire is a Likert-type questionnaire consisting of 10 items and two sub-dimensions, "progression" and "obstruction". Progress sub-dimension emphasized being able to do daily tasks in line with values, while blocking sub-dimension emphasized living a life away from values in activities carried out for a week, unlike progress. The Cronbach's alpha value for the whole scale is 0.78. The lowest total score is zero, while the highest is 60. A high score indicates that individuals live a life in line with their values

CONTACTS AND LOCATIONS:
Overall Officials: Elif C Bulut, Msc, Principal Investigator — Dokuz Eylul University; Elif can Bulut, Msc, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338